CLINICAL TRIAL: NCT02886299
Title: Comparative Study of Effects and Safety of Intermittent Low Dose Therapy of Fenofibrate and Simvastatin on Chronic Hemodialysis Patients
Brief Title: Randomized Comparative Efficacy and Safety Study of Intermittent Simvastatin and Fenofibrate in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohammed Abdel Magid Abdel Hamid, Teaching Assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL (746)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Fenofibrate/Simvastatin Comparison
Keywords: Fibrates; Statins; Hemodialysis; Dyslipidemia; Improved Oxidative Stress; Egypt
MeSH Terms: conditions — Dyslipidemias | interventions — Fenofibrate; Simvastatin

ARMS (2):
- Fenofibrate group (Active Comparator): Group I (30 patients): Patients receiving fenofibrate (100 mg) taken on dialysis days after the dialysis session (three times per week).
  Interventions: Drug: Fenofibrate
- Simvastatin group (Active Comparator): Group II (30 patients): Patients receiving simvastatin (20 mg) taken on dialysis days after the dialysis session (3 times per week).
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Fenofibrate
  Arms: Fenofibrate group
Drug: Simvastatin
  Arms: Simvastatin group

SUMMARY:
Sixty chronic hemodialysis patients were randomly assigned to receive fenofibrate 100 mg (group 1, n = 30) or simvastatin 20 mg (group 2, n = 30) three times/week after their dialysis session. The safety and efficacy of drugs on lipid profile, oxidized low density lipoproteins (ox-LDL), glutathione peroxidase (GSH-Px) and C-reactive protein (CRP) were compared before and after 16-week treatment.

DETAILED DESCRIPTION:
This is a prospective randomized open label parallel study.

The selected patients will be randomly allocated to one of two groups

* Group I (30 patients): Patients receiving fenofibrate (100 mg) taken on dialysis days after the dialysis session (three times per week).
* Group II (30 patients): Patients receiving simvastatin (20 mg) taken on dialysis days after the dialysis session (3 times per week).

A careful history of all patients including demographic characteristics, physical examination, chief complaint, past medical history, drug history, familial history, social history, disease(s).

Monitoring Parameters:

For efficacy, the following parameters are measured:

1. Lipid profile (total cholesterol, HDL, TG and LDL from Friedwald formula [10] {LDL-C= TC-[HDL + TG\5]). (measured at baseline and every month for 4 months)
2. C-reactive protein (CRP). (measured at baseline and after 4 months)
3. Oxidative stress markers: oxidized LDL and human glutathione peroxidase (measured at baseline and after 4 months).

For safety: (measured at baseline and every month for 4 months)

1. Observe for signs & symptoms of muscle toxicity and measure phosphocreatine kinase (CPK).
2. Liver function tests: ALT, AST, ALP & albumin.
3. Urea & serum creatinine. (to monitor renal function)
4. Hemoglobin
5. Other measurements: Body mass index (BMI), Blood Pressure, electrolytes (Sodium,potassium, calcium, phosphorous) and assess patient compliance by tablet counting.

Statistical analysis will be used to compare the effects of simvastatin and fenofibrate on lipid profile, inflammatory marker (CRP) and oxidative stress markers (oxidized LDL and glutathione peroxidase). In addition, comparing their safety on renal and hepatic functions, phosphocreatine kinase, blood pressure and blood glucose level.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Chronic hemodialysis patients with 3 dialysis sessions per week.
3. Lipid profile:

   1. Total Cholesterol ≥ 200 mg/dl or LDL ≥ 130 mg/dl.
   2. Triglycerides ≥ 150 mg/dl.

Exclusion Criteria:

1. Previous intolerance to fibrates or statins.
2. Use of any fibrates or statins within 6 months prior to study.
3. Hypothyroidism.
4. Active liver disease [unexplained persistent increase in liver enzymes (ALT & AST > 2x ULN)].
5. Uncontrolled hypertension.
6. History of MI or coronary bypass surgery in last 3 months.
7. Muscle toxicity (Phosphocreatine kinase (CPK) > 2x ULN).
8. Gall bladder disease.
9. Use of any immunosuppressant or steroid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
oxidative stress markers (serum ox-LDL and GSH-Px) | 16 weeks
C-reactive protein | 16 weeks